CLINICAL TRIAL: NCT05430360
Title: Single-center, Single-arm Phase I Clinical Study of Autologous Tumor-infiltrating Lymphocyte Injection (GT201) for the Treatment of Metastatic/recurrent Advanced Solid Tumors
Brief Title: Autologous Tumor-infiltrating Lymphocyte Injection (GT201) for the Treatment of Metastatic/recurrent Advanced Solid Tumors
Acronym: GT201
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CO-FA-018
Record Dates: First submitted 2022-06-04; First posted 2022-06-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT201 treatment group (Experimental): Autologous tumor infiltrating lymphocyte injection
  Interventions: Biological: GT201

INTERVENTIONS:
Biological: GT201 — Autologous tumor infiltrating lymphocyte injection

SUMMARY:
This study is a single-center, single-arm phase I clinical trial. A total of 30 subjects (20 evaluable cases are expected) from 1 cohort will be enrolled in this study.

An "autologous tumor-infiltrating lymphocyte therapy" dosing regimen consisting of lymphodepleting chemotherapy (FC regimen: cyclophosphamide + fludarabine), infusion of autologous tumor-infiltrating lymphocyte injection, and interleukin-2 injection will be used.The study process is divided into: screening period, sampling and production period, clearing and chemotherapy period, treatment and observation period, and follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily enrolled in the study, signed an informed consent form, and willing and able to comply with the study protocol
2. At least one lesion (preferably superficial lymph nodes) that has not been treated with radiation, has not received other local therapies, has access to tumor tissue, and can isolate at least a mass ≥ 1.0 g of tissue mass (either single lesion source or multiple lesions combined) for the preparation of autologous tumor-infiltrating lymphocytes
3. Eastern Collaborative Oncology Group (ECOG) physical fitness status score of 0 or 1.

Exclusion Criteria:

1. Failure of surgery and/or radiation therapy to relieve spinal cord compression is not eligible for enrollment
2. People with uncontrolled tumor-related pain as judged by the investigator
3. Risk of major bleeding as assessed by investigators
4. Have interstitial pneumonia or clinically significant active pneumonia at screening, or other respiratory disease that severely affects lung function
5. Any active autoimmune disease 14 days prior to clear lymphatic chemotherapy, history of autoimmune disease, or disease requiring systemic steroid hormone or immunosuppressive drug therapy 6:History of allergic reaction to any component of the drugs to be used in the study (including but not limited to autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, interleukin-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40, antibiotics (beta-lactam antibiotics, gentamicin));

7：Women who are pregnant or breastfeeding; or women who are pregnant, breastfeeding, or planning to become pregnant within 1 year of the cell return.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adcersed events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection（GT201) in patients with relapsed/metastatic advanced solid tumor as measured by the incidence and severity of adcersed events per CTCAE 5.0

SECONDARY OUTCOMES:
Objective response rate | 3 years
  To evaluate efficacy parameters such Objective Response Rate (ORR) per RECIST 1.1, as assessed by the Investigator
Progression-free survival | 3 years
  To evaluate efficacy parameters such Progression-Free Survival (PFS) per RECIST 1.1, as assessed by the Investigator
Overall survival | 3 years
  To evaluate efficacy parameters such Overall Survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No